CLINICAL TRIAL: NCT03106545
Title: Ultrasound-guided Specific Blocks of the Distal Tibial and Deep Peroneal Nerves at the Level of the Ankle With a Mixture of Bupivacaine + Liposome Bupivacaine v Bupivacaine Alone v General Anesthesia
Brief Title: Liposome Bupivacaine for ANKLE Blocks
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catherine Vandepitte, M.D. (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor-Investigator, Catherine Vandepitte, M.D., Director, New York School of Regional Anesthesia
Organization: New York School of Regional Anesthesia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1602
Record Dates: First submitted 2017-03-24; First posted 2017-04-10 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Hallux Valgus (Bunions)
MeSH Terms: conditions — Hallux Valgus; Bunion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single mixture LB & bupivacaine (Experimental): A single mixture of liposome bupivacaine 1.3% (5 mL) + bupivacaine 0.5% (2.5 mL) injected into the distal tibial and deep peroneal nerves
  Interventions: Drug: Liposome bupivacaine
- Bupivacaine alone (Active Comparator): Bupivacaine 0.5% (7.5 mL) injected into the distal tibial and deep peroneal nerves
  Interventions: Drug: Liposome bupivacaine
- General anesthesia (Sham Comparator): General anesthesia
  Interventions: Drug: Liposome bupivacaine

INTERVENTIONS:
Drug: Liposome bupivacaine

SUMMARY:
Postoperative analgesia for hallux valgus surgery (bunionectomy) is inconsistent and may even result in rebound pain when the (ankle) blocks wear off. It is hypothesized that the mixture of bupivacaine and liposome bupivacaine increases the extent and duration of postoperative analgesia and decreases opioid consumption as compared to bupivacaine alone or to general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years and max 65 years of age at screening
* Scheduled to undergo primary Scarf osteotomy for elective hallux valgus
* American Society of Anesthesiologists (ASA) physical status 1, 2, or 3
* Female subject must be surgically sterile or have a monogamous partner who is surgically sterile; or be at least 2 years postmenopausal; or practicing abstinence; or using an insertable, injectable, transdermal, or combination oral contraceptive approved by the FDA for greater than 2 months prior to screening and commit to the use of an acceptable form of birth control for the duration of the study and for 30 days after completion of the study
* Able to demonstrate sensory function by exhibiting sensitivity to cold, pinprick, and light touch
* Able to understand the English or Dutch language, purpose and risks of the study, provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations
* Able to adhere to the study visit schedule, and complete all study assessments.

Exclusion Criteria:

* Currently pregnant, nursing, or planning to become pregnant during the study or within 1 month after study drug administration
* Planned concurrent surgical procedure (e.g., bilateral hallux valgus repair)
* Concurrent painful physical condition that may require analgesic treatment (such as an NSAID or opioid) in the postsurgical period for pain that is not strictly related to hallux valgus and which may confound the postsurgical assessments (e.g., significant pain from other joints including chronic neuropathic pain, concurrent or prior contralateral knee or foot surgery)
* Previous hallux valgus on the foot being considered for surgery
* History of hypersensitivity or idiosyncratic reaction to amide-type local anesthetics
* Contraindication to bupivacaine, oxycodone, morphine, or hydromorphone
* Chronic daily use of long-acting opioid medication or NSAIDs (except for low-dose aspirin used for cardioprotection) within 24 hours
* Initiation of treatment with any of the following medications within 1 month of study drug administration or if the medication(s) are being given to control pain: selective serotonin reuptake inhibitors (SSRIs), selective norepinephrine reuptake inhibitors (SNRIs), gabapentin, pregabalin (Lyrica®), or duloxetine (Cymbalta®). If a subject is taking one of these medications for a reason other than pain control, he or she must be on a stable dose for at least 1 month prior to study drug administration.
* Current use of systemic glucocorticosteroids within 1 month of study enrollment
* Use of dexmedetomidine HCl (Precedex®) within 3 days of study drug administration
* History of impaired kidney function, chronic respiratory disease, rheumatoid arthritis, coagulopathy, or loss of sensation in the extremities
* Impaired kidney function (e.g., serum creatinine level >2 mg/dL [176.8 µmol/L] or blood urea nitrogen level >50 mg/dL [17.9 mmol/L]) or impaired liver function (e.g., serum aspartate aminotransferase [AST] level >3 times the upper limit of normal (ULN) or serum alanine aminotransferase [ALT] level >3 times the ULN
* Uncontrolled anxiety, psychiatric, or neurological disorder that might interfere with study assessments
* Any chronic neuromuscular deficit affecting the peripheral nerves or muscles of the surgical extremity
* Any chronic condition or disease that would compromise neurological or vascular assessments
* Suspected or known history of drug or alcohol abuse within the previous year
* Body weight <40 kg (88 pounds) or a body mass index >44 kg/m2
* Previous participation in an EXPAREL study
* Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Change in current pain over the first postoperative week | From baseline (before nerve block) through first postoperative week
  Pain rating (NRS) at rest and with movement
Change in worst pain over the first postoperative week | From discharge from PACU through first postoperative week
  Modified BRIEF Pain Inventory (Q1)

SECONDARY OUTCOMES:
Opioid consumption | From hospital discharge through first postoperative week
  Self-reported consumption of Tramadol tablets
Change in ability to use foot | From discharge from PACU through first postoperative week
  Stand with equal weight on both feet, wiggle toes, walk 10 steps
Change in sleep quality | From discharge from PACU through first postoperative week
  Duration (h), quality rating (0 - 10)
Change in satisfaction with pain control | From discharge from PACU through first postoperative week
  With pain control (0 - 10)
Change in sensory response in skin dermatomes | From premedication through first postoperative week
  Cold, pinprick, light touch in the distal tibial and deep peroneal nerve dermatomes
Change in motor response in foot | From premedication through first postoperative week
  Plantar flexion, dorsiflexion

OTHER OUTCOMES:
Total number of participants with side effects to regional anesthesia peripheral nerve blockade | From beginning of nerve block through first postoperative week
  Nausea, vomiting, fever, constipation, severe itching of the skin, dizziness, sleepless nights, excessive sweating, urinary retention, headache, heart palpitations
Participants with adverse events | From date of signing ICF through first postoperative week
  Any untoward medical occurrence (unfavorable and/or unintended change in a body structure or body function) associated with the use of a drug in humans, whether or not considered drug related

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: No